CLINICAL TRIAL: NCT04696133
Title: Therapeutic Outcomes of Sensory Integration Versus Fine Motor Intervention on Autistic Features and Fine Motor Skills in Children With Autism: A Randomized Controlled Trial
Brief Title: Sensory Integration Versus Fine Motor Intervention in Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Mahmoud Abd-elmonem, Amira Abd-elmonem, assist Prof. Physiacl therapy for pediatric department, faculty of physical therapy , Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Autism spectrum
Record Dates: First submitted 2021-01-03; First posted 2021-01-06 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Quality of life; sensory integration; fine motor skills
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional training (Experimental): children received fine motor exercises
  Interventions: Other: fine motor skills
- sensory integration training (Experimental): Children received designed sensory integration program
  Interventions: Other: sensory integration

INTERVENTIONS:
Other: fine motor skills — stretching and strengthening exercises in addition to exercises to enhance fine motor skills
  Arms: conventional training
Other: sensory integration — * Tactile stimulation
  * Proprioceptive stimulation
  Arms: sensory integration training

SUMMARY:
Clinically, infants with Autism spectrum often display gross motor delays in supine, prone, and sitting skills in their first year of life.

ELIGIBILITY:
Inclusion Criteria:

* Age ranges from 8 to 12 years.
* Mild to moderate autistic features

Exclusion Criteria:

• Significant visual or auditory defects.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Gilliam autism rating scale | 3 months
  higher the autism index, indicate the probability the individual has autism

SECONDARY OUTCOMES:
Bruininks-Oseretsky Test Of Motor Proficiency | 3 months
  Fine manual control domain will be assessed in the current study. Gender specific norms were used for scoring as the scale's authors report these as being more accurate than combined gender norms

CONTACTS AND LOCATIONS:
Overall Officials: Emam H El-Negamy, professor, Study Chair — Cairo University; kamilia saad, Study Director — Cairo University; dalia galal, Principal Investigator — Cairo university, Egypt
Locations (1):
- faculty of physical therapy, Cairo university, Giza, Egypt